CLINICAL TRIAL: NCT07352124
Title: Rosemary Infusion for Hypertension With Hypertriglyceridemia: A Triglyceride-Stratified Clinical Study
Brief Title: Rosemary Infusion for Hypertension With Hypertriglyceridemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: awatef Sassi (Other)
Responsible Party: Sponsor-Investigator, awatef Sassi, Laboratory of Cardiopulmonary System Interactions, Faculty of Medicine, Sousse
Organization: Faculty of Medicine, Sousse (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TGhypertension
Record Dates: First submitted 2026-01-11; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Hypertension With Hypertriglyceridemia
Keywords: Rosemary infusion, hypertension , Hypertriglyceridemia
MeSH Terms: conditions — Hypertension; Hypertriglyceridemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Groupe triglycérides normaux TG < 1,7 mmol/L n = 22 (Experimental)
  Interventions: Dietary Supplement: Rosemary infusion
- TG ≥ 1,7 mmol/L n = 25 (Experimental)
  Interventions: Dietary Supplement: rosemary infusion

INTERVENTIONS:
Dietary Supplement: Rosemary infusion — Rosemary infusion 100 ml during 45 days
  Arms: Groupe triglycérides normaux TG < 1,7 mmol/L n = 22
Dietary Supplement: rosemary infusion — Rosemary infusion 100 ml during 45 days
  Arms: TG ≥ 1,7 mmol/L n = 25

SUMMARY:
This study aimed to evaluate the effects of daily rosemary infusion consumption on blood pressure and lipid profile in patients with mild hypertension, stratified by triglyceride status.

This 6-week open-label interventional study enrolled 47 patients with mild hypertension (systolic BP 140-159 mmHg and/or diastolic BP 90-99 mmHg). Participants were stratified into two groups: normal triglycerides, TG <1.7 mmol/L, n=22 and high triglycerides, TG ≥1.7 mmol/L, n=25. Blood pressure was assessed using 24-hour ambulatory monitoring (Holter) at baseline and day 45. Comprehensive biochemical analysis included lipid profile, hepatic and renal function markers, and inflammatory parameters.

ELIGIBILITY:
Inclusion Criteria:

Participants of both sexes, aged 18 years and older, were included in the study. The inclusion criteria were: (1) Presence of mild hypertension defined as systolic blood pressure (SBP) of 140-159 mmHg and/or diastolic blood pressure (DBP) of 90-99 mmHg according to the 2018 ESC/ESH guidelines(Williams et al., 2018); (2) No use of medications or dietary supplements for other health conditions.

Exclusion Criteria:

Participants were excluded if they had renal failure, autoimmune diseases, major gastrointestinal disorders, or a history of cardiovascular disease. Other exclusion criteria included current or past use of medications known or suspected to influence blood pressure or metabolic parameters

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Blood pressure measurement | 45 days
Evolution of serum triglycerides | 45 days

SECONDARY OUTCOMES:
Cardiovascular disease risk assessment | 45 days
Atherogenic Index of Plasma | 45 days

CONTACTS AND LOCATIONS:
Locations (1):
- Sassi, Sousse, Tunisia

IPD SHARING:
Plan to Share IPD: No